CLINICAL TRIAL: NCT05248555
Title: The National Australian HCV Point-of-Care Testing Program: An Observational Cohort Study to Evaluate the Use of Finger-stick Point-of-care Hepatitis C Testing to Enhance Diagnosis and Treatment of HCV Infection - Minimal Dataset
Brief Title: The National Australian HCV Point-of-Care Testing Program - Minimal Dataset
Status: Recruiting | Type: Observational
Sponsor: Kirby Institute (Other Government)
Collaborators: Flinders University (Other)
Responsible Party: Sponsor
Other Study IDs: VHCRP2104
Record Dates: First submitted 2021-12-12; First posted 2022-02-21 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Hepatitis C
Keywords: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People at risk of HCV acquisition: Clinic staff will offer HCV point-of-care testing to participants as they access services. Testing will be performed using point-of-care HCV RNA testing.
  Interventions: Diagnostic Test: Point-of-Care Testing

INTERVENTIONS:
Diagnostic Test: Point-of-Care Testing — Participants will be offered finger-stick point-of-care testing for HCV

SUMMARY:
The National Australian HCV Point-of-Care Testing Program will establish an observational cohort to evaluate whether scale-up of finger-stick point-of-care HCV testing increases diagnosis and treatment for HCV infection. Participants will be recruited from settings providing services to people with a risk factor for the acquisition of HCV infection (including drug treatment clinics, needle and syringe programs, homelessness settings, mental health services, prisons, and mobile outreach). All participants who undergo HCV point-of-care testing at the study site will be included in the data collection. Participants will not receive treatment as a part of this study. Participants who are HCV RNA positive will be linked to standard of care.

DETAILED DESCRIPTION:
The advent of simple direct-acting antiviral hepatitis C (HCV) therapies with cure rates >95% is one of the greatest medical advances in decades, having led to a reversal in liver-related mortality. In Australia, treatment uptake has declined between 2016 (32,000 treated) and 2019/20 (2019: 11,500; 2020: 8,500).1 Progress towards HCV elimination has been impeded by COVID-19, affecting the delivery of national and state-based HCV strategies. Improving HCV treatment uptake to reduce disease burden is a key aim of global, national and state-based HCV strategies.2-4

Scale-up of HCV testing and treatment will be required to achieve elimination by 2030. Current diagnostic pathways require multiple visits to a practitioner reducing the proportion who receive a diagnosis. In Australia, 81% of people have had HCV antibody testing (indicates exposure), but only 47% have been HCV RNA tested (indicates active infection and the need for HCV treatment).5 Mathematical modelling suggests that HCV RNA testing needs to increase by at least 50% annually to achieve elimination in Australia by 2030.6

The Kirby Institute is an international leader in research evaluating the Xpert HCV assay (Grebely Lancet Gastro Hep 2017), having built a large network of Xpert platforms for HCV testing in needle and syringe programs, prisons, drug treatment clinics, tertiary hospitals, and Aboriginal Community Controlled Health Service. In Kirby-led research, point-of-care HCV testing interventions in needle and syringe programs and prisons have resulted in high HCV treatment uptake (70-90%). The Kirby Institute and Flinders University also have a strong track record of implementing point-of-care testing for STIs and COVID-19, providing an ideal foundation to scale-up Xpert HCV testing in Australia.

The Kirby Institute and Flinders University will establish the Australian National HCV Point-of-care Testing Program for the scale-up of point-of-care HCV RNA testing in services with high prevalence of HCV infection, including community health centres, drug treatment clinics, needle and syringe programs, and prisons. This program will include the development of standard operating procedures, logistics/deployment, initial set-up, an operator training program, and quality assurance and competency assessment program.

An observational cohort study will be established to evaluate HCV treatment uptake following scale-up of point-of-care HCV testing among people with a risk factor for acquisition of HCV infection or people attending a service caring for people with risk factors for the acquisition of HCV infection.

Participants will be recruited from settings that provide services to people with a risk factor for the acquisition of HCV infection. All participants who undergo point-of-care HCV testing at the study site will be included in the data collection. Participants will not receive treatment as a part of this study. Participants who are HCV RNA positive will be linked to standard of care for any other clinical assessments and treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Received point-of-care HCV testing.

Exclusion Criteria:

* Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from settings that provide services to people with a risk factor for the acquisition of HCV infection, including drug treatment clinics, needle and syringe programs, prisons, mobile outreach services, community health services, mental health services, homelessness services, and other appropriate settings nationally. It is anticipated approximately 40,000 participants will be screened for HCV infection using point-of-care HCV testing.
Sampling Method: Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of HCV infected participants who initiate HCV treatment at 12 weeks | 12 Weeks from enrolment
  To evaluate the proportion of HCV infected (HCV RNA quantifiable) participants who initiate HCV treatment at 12 weeks following finger-stick point-of-care HCV RNA testing.

SECONDARY OUTCOMES:
The proportion of participants who accept point-of-care testing | 2 years from recruitment commencement
  To evaluate the proportion of people who accept point-of-care testing among those offered testing.
The prevalence of HCV infection amongst study participants tested | 2 years from recruitment commencement
  To evaluate the prevalence of current HCV infection (HCV RNA quantifiable) among people tested.
To evaluate the time to HCV treatment uptake among HCV RNA positive participants | 52 weeks
  To evaluate the length of time participants take to initiate HCV treatment after diagnosis
To evaluate proportion of HCV RNA positive participants who initiate HCV treatment | 52 weeks
  To evaluate the proportion of HCV RNA positive participants who initiate HCV treatment at 12 months (52 weeks) following finger-stick point-of-care HCV RNA testing.
To evaluate the proportion of participants who complete HCV (DAA) treatment | 52 weeks
  To evaluate the proportion of participants who complete HCV direct-acting antiviral (DAA) treatment.
To evaluate the proportion of participants who achieve an SVR | 12 weeks
  To evaluate the proportion of participants who achieve an SVR (defined as HCV RNA below the lower limit of quantitation at post treatment week 12).
To evaluate the proportion of participants who are HCV RNA negative at 12 months | 52 weeks
  To evaluate the proportion of participants who are HCV RNA negative at 12 months (52 weeks) following finger-stick point-of-care HCV RNA testing.

CONTACTS AND LOCATIONS:
Locations (11):
- Australia (11):
  - Justice Health and Forensic Mental Health Network, Sydney, New South Wales
  - Lotus Glen Correctional Centre, Cairns, Queensland
  - Hepatitis Queensland, Coorparoo, Queensland
  - West Moreton Hospital and Health Service, Ipswich, Queensland
  - Townsville Correctional Centre, Townsville, Queensland
  - Woodford Correctional Centre, Woodford, Queensland
  - South Australian Prison Health Service, Marden, South Australia
  - Mount Gambier Priosn, Mount Gambier, South Australia
  - St Vincent's Correctional Health Services, Fitzroy, Victoria
  - Medically Supervised Injecting Room, Melbourne, Victoria
  - Geo Healthcare - The Geo Group Australia Pty Ltd, Ravenhall, Victoria